CLINICAL TRIAL: NCT03407313
Title: The CONFORM Study: A Multi-center Study to Evaluate the Safety and Efficacy of Rotational Fractional Resection on Submental Contouring
Brief Title: CONFORM: Rotational Fractional Resection for Submental Contouring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recros Medica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-0002
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Skin Laxity; Lipodystrophy
Keywords: Submental fullness; Submental fat; Loose skin
MeSH Terms: conditions — Cutis Laxa; Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Rotational fractional resection (1.5mm diameter device) (Experimental): Single treatment of skin resection and focal lipectomy (removal of loose skin and fat)
  Interventions: Device: Rotational fractional resection (1.5mm diameter device)

INTERVENTIONS:
Device: Rotational fractional resection (1.5mm diameter device) — Single treatment of skin resection and focal lipectomy (removal of loose skin and fat)

SUMMARY:
This study will evaluate the safety and efficacy of rotational fractional resection (RFR) to improve neck contouring. RFR is used to remove loose skin and fat.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm (non-randomized), interventional cohort, non-significant risk (NSR) study designed to investigate the efficacy and safety of Rotational Fractional Resection (skin resection and focal lipectomy) in patients with mild to moderate submental fat and mild to moderate submental skin laxity. The total duration of study participation for each subject is approximately up to 7 months for each subject from the screening visit to the exit visit. The follow-up period will be approximately 6 months after the procedure. Eligible subjects will complete a total of 8 study visits: screening, procedure, and follow-up visits at 1, 7, 14, 30, 90 and 180 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, at least 30 years old
* Moderate submental (neck) fat
* Mild to moderate submental (neck) skin laxity (loose skin)
* Willing and able to provide informed consent
* Willing and able to comply with all protocol requirements
* Willing to limit direct sun exposure and use sunscreen for duration of the study
* Agree to maintain weight for duration of the study
* Willing to have photographs taken that could identify the participant

Exclusion Criteria:

* Previous intervention to treat submental fat or skin laxity
* Use of aspirin, ibuprofen, naproxen, or Vitamin E within 14 days of the procedure
* Sensitivity to local anesthesia
* Severe acne, cystic acne or acne scars on neck
* Trauma of chin or neck area
* Skin infection or rash on neck
* Psoriasis, eczema, rosacea, or vitiligo
* History of scarring
* History or current symptoms of dysphagia
* Chronic or persistent coughing
* Body mass index (BMI) > 30
* Clinically significant bleeding disorder
* Anemia, kidney disease, or liver disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Knowlton, MD, Study Director — Recros Medica, Inc.
Locations (6):
- United States (6):
  - Aesthetx, Campbell, California
  - Steve Yoelin, MD Medical Associates, Inc., Newport Beach, California
  - Roseville Facial Plastic Surgery, Roseville, California
  - Miami Dermatology & Laser Institute, Miami, Florida
  - DeNova Research, Chicago, Illinois
  - Sundaram Dermatology, Cosmetic & Laser Surgery Center, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rotational Fractional Resection (1.5mm Diameter Device): Single treatment of skin resection and focal lipectomy (removal of loose skin and fat) in submentum
Period: Overall Study
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Started | 68
Completed | 66
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 67
  More than one race | 1
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.7 (3.1)
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type (Grades I through IV) is a numerical classification schema for human skin color
  Participants
    Type I - Ivory white (pale white); extremely fair skin | 2
    Type II - White or fair skin | 36
    Type III - Medium white skin | 30
    Type IV - Beige or lightly tanned or olive skin | 0
    Type V - Moderately brown or tanned brown skin | 0
    Type VI - Dark brown or black skin | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction of Submental Skin Area ≥ 20 mm^2
Description: This endpoint is the difference in the measurement of submental skin area (mm^2) between Baseline and 90 days. A reduction of ≥ 20 mm^2 denotes improvement.
Time Frame: Baseline and 90 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Number analyzed (Participants) | 68
Participants | 49

2. Secondary Outcome: Number of Participants Who Were Satisfied With the Appearance of Their Neck and Jawline
Description: Subjects rated their satisfaction of the appearance of their neck and jawline on a Subject Satisfaction Questionnaire. Results reflect subjects who were satisfied ("somewhat satisfied", "satisfied", or "very satisfied").
Time Frame: 90 days after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Number analyzed (Participants) | 68
Participants | 56

3. Secondary Outcome: Number of Participants With Post-treatment Images Correctly Identified
Description: Correct identification of post-treatment images by three blinded independent reviewers in more than 50% of subjects
Time Frame: Pre-treatment and 90 days after treatment
Population: 68 subjects were assessed by three blinded reviewers
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
Number analyzed (Participants) | 68
Participants
  Blinded Reviewer 1 | 59
  Blinded Reviewer 2 | 67
  Blinded Reviewer 3 | 67

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Rotational Fractional Resection (1.5mm Diameter Device)
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 45/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotational Fractional Resection (1.5mm Diameter Device) (N=68)
Administration site erythema (Injury, poisoning and procedural complications) | 11
Administration site bruising (Injury, poisoning and procedural complications) | 11
Contact Dermatitis (Injury, poisoning and procedural complications) | 4
Hypoaesthesia (Injury, poisoning and procedural complications) | 4
Skin Mass (Skin and subcutaneous tissue disorders) | 5
Abnormal Skin Texture (Injury, poisoning and procedural complications) | 6
Nausea (Gastrointestinal disorders) | 4

LIMITATIONS AND CAVEATS:
This study evaluated 1.5mm diameter skin resections, our first-generation prototype, in the submentum area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT03407313/Prot_SAP_000.pdf